CLINICAL TRIAL: NCT02263937
Title: Double Blind, Randomised, Dual Centre, Crossover, Pilot Trial of Bilateral Nucleus Basalis of Meynert Deep Brain Stimulation to Improve Cognitive Deficits in Patients With Dementia With Lewy Bodies.
Brief Title: Deep Brain Stimulation for Patients With Dementia With Lewy Bodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13/0538
Record Dates: First submitted 2014-09-30; First posted 2014-10-13 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilateral Nucleus Basalis Meynert DBS (Active Comparator): 6 week period of active NBM DBS
  Interventions: Procedure: Bilateral Nucleus Basalis Meynert DBS
- Sham Nucleus Basalis Meynert DBS (Sham Comparator): 6 week period of Sham DBS
  Interventions: Procedure: Sham Nucleus Basalis Meynert DBS

INTERVENTIONS:
Procedure: Bilateral Nucleus Basalis Meynert DBS — Low frequency stimulation applied using standard Deep brain stimualtion hardware.
  Other Names: Active Deep Brain Stimulation
  Arms: Bilateral Nucleus Basalis Meynert DBS
Procedure: Sham Nucleus Basalis Meynert DBS — DBS system switched off.
  Other Names: Sham DBS
  Arms: Sham Nucleus Basalis Meynert DBS

SUMMARY:
This trial aims to collect pilot data to explore whether bilateral deep brain stimulation (DBS) of the Nucleus Basalis of Meynert (NBM) has beneficial effects on memory and thinking impairments among individuals with Dementia with Lewy Bodies (DLB).

DETAILED DESCRIPTION:
We will perform a pilot study to evaluate the effectiveness of human NBM DBS at improving cognitive deficits in DLB patients. Six patients with DLB with moderate cognitive impairments (including but not restricted to deficits in attention and working memory) will have bilateral DBS electrodes implanted to ensure that superficial contacts lie in the motor Globus Pallidum interna (GPi) target, while the deepest electrical contacts lie in the NBM. We will place electrodes using our conventional image-guided, stereotactic frame-based procedure. Once the surgical wounds have healed, patients will be randomised into 2 groups in a crossover trial design to have 6 week periods of NBM stimulation switched on or switched off separated by a 2 week washout period, following which the patient will cross over to have the opposite condition for a further 6 weeks. Outcome measures collected at the 6 weeks and 14 weeks timepoints will be compared according to whether each patient was ON or OFF stimulation at that timepoint.

At the end of the crossover period, all patients will be invited for continued follow up with stimulation switched on and will have neuropsychological evaluations at 6 monthly intervals. Patients will be given the option of receiving additional conventional stimulation to the motor GPi, through the higher contacts of each electrode, at the end of the crossover period if required for any coexisting Parkinsonian motor complications of DLB.

ELIGIBILITY:
Inclusion Criteria:

* DLB Consortium Criteria for diagnosis
* Score between 2 & 12 on Clinician Assessment of Fluctuations scale
* MMSE score between 21 and 27
* Appropriate Surgical candidates in terms of general health
* Aged between 50 & 80
* Able to give Informed consent
* Living at home with Carer
* Able to comply with protocol
* On stable dosage of cholinesterase inhibitor

Exclusion Criteria:

* Diagnosis of other cause for dementia
* Abnormality on brain imaging considered likely to compromise compliance with trial protocol.
* Prior intracerebral surgical intervention

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Hopkins Verbal Learning test | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Verbal Fluency | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Simple & Choice Reaction time task | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Wechsler Adult Intelligence scale (WAIS IV) Digit Span | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Posner's Covert Attention test | Comparing ON v OFF at 6 weeks & 14 weeks according to stimulation status
Clinician's Assessment of Fluctuations scale | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status

SECONDARY OUTCOMES:
Minimental State Examination (MMSE) | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Dementia Rating Scale (DRS-2) | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Wechsler Abbreviated Scale of Intelligence (WASI) | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Short Recognition Memory | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Wechsler Adult Intelligence Scale IV -Letter, Number sequencing | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Trail Making test | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Stroop test | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Wechsler Adult Intelligence Scale IV - Symbol search | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Judgement of Line Orientation | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
North East Visual Hallucinations Interview | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Neuropsychiatric Inventory | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Florida Apraxia Screening test | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Clinical Global Impression Scale | Comparing ON v OFF at 6 weeks & 14 weeks according to stimulation status
Hamilton Depression scale | Comparing ON v OFF at 6 weeks & 14 weeks according to stimulation status
Hamilton Anxiety Scale | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Starkstein Apathy Rating scale | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Movement Disorders Society- Unified Parkinson's Disease Rating Scale | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Freezing of Gait- questionnaire | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Scales for outcome in Parkinson's disease (SCOPA - AUT) | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Quality of Life- Alzheimer's Disease | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Mayo Fluctuations Composite Scale | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Blessed Dementia scale | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Carer Strain Index | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status
Short Form 36 | Comparing ON v OFF stimulation at 6 weeks & 14 weeks according to stimulation status

OTHER OUTCOMES:
Adverse Events | Throughout trial period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Foltynie, MB BS MRCP, Principal Investigator — UCL Institute of Neurology
Locations (2):
- United Kingdom (2):
  - UCL Institute of Neurology, London
  - University of Newcastle, Newcastle

REFERENCES:
- [Derived] Gratwicke J, Zrinzo L, Kahan J, Peters A, Brechany U, McNichol A, Beigi M, Akram H, Hyam J, Oswal A, Day B, Mancini L, Thornton J, Yousry T, Crutch SJ, Taylor JP, McKeith I, Rochester L, Schott JM, Limousin P, Burn D, Rossor MN, Hariz M, Jahanshahi M, Foltynie T. Bilateral nucleus basalis of Meynert deep brain stimulation for dementia with Lewy bodies: A randomised clinical trial. Brain Stimul. 2020 Jul-Aug;13(4):1031-1039. doi: 10.1016/j.brs.2020.04.010. Epub 2020 Apr 22. PMID 32334074